CLINICAL TRIAL: NCT05444257
Title: A Phase 3, Open-label Study Evaluating the Long-term Safety and Efficacy of VX-121/TEZ/D-IVA Combination Therapy in Subjects With Cystic Fibrosis
Brief Title: A Study Evaluating the Long-term Safety and Efficacy of VX-121 Combination Therapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX20-121-104; 2021-000713-17 (EudraCT Number); 2024-514173-22-00 (Other: EU CT Number)
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VX-121/TEZ/D-IVA (Experimental): Part A: Participants will receive VX-121/TEZ/D-IVA once daily for 96 weeks. Part B: Participants will receive VX-121/TEZ/D-IVA once daily for an additional 48 weeks.
  Interventions: Drug: VX-121/TEZ/D-IVA

INTERVENTIONS:
Drug: VX-121/TEZ/D-IVA — Fixed-dose combination tablets for oral administration.
  Other Names: VX-121/VX-661/CTP-656; VX-121/VX-661/VX-561; VX-121/tezacaftor/deutivacaftor

SUMMARY:
The purpose of this study is to evaluate the long-term safety, tolerability, and efficacy of VX-121/tezacaftor/deutivacaftor (VX-121/TEZ/D-IVA) in participants with cystic fibrosis.

ELIGIBILITY:
Key Inclusion Criteria:

* Part A: Completed study drug treatment in a parent study VX20-121-102 (NCT05033080) and VX20-121-103 (NCT05076149); or had study drug interruption(s) in a parent study but did not permanently discontinue study drug, and completed study visits up to the last scheduled visit of the Treatment Period in the parent study
* Part B: Completed study drug treatment in Part A; or had study drug interruption(s) in Part A, but did not permanently discontinue study drug, and completed study visits up to the last scheduled visit of the Treatment Period of Part A

Key Exclusion Criteria:

* History of drug intolerance in a parent study
* Pregnant or breast-feeding females at the time of enrollment in Part A

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 822 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Baseline up to Week 148

SECONDARY OUTCOMES:
Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) | From Baseline up to Week 144
Absolute Change From Baseline in Sweat Chloride (SwCl) | From Baseline up to Week 144
Number of Pulmonary Exacerbations (PEx) | From Baseline up to Week 144

CONTACTS AND LOCATIONS:
Locations (195):
- United States (72):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Miller Children's Hospital / Long Beach Memorial, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente, Oakland, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California San Francisco, Lung Transplant Program, San Francisco, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - University of Florida, Shands Hospital, Gainesville, Florida
  - Joe DiMaggio Cystic Fibrosis & Pulmonary Center, Hollywood, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Central Florida Pulmonary Group,PA, Orlando, Florida
  - Nemours Children's Specialty Care, Pensacola, Florida
  - Johns Hopkins All Children's Hospital Outpatient Care Center, St. Petersburg, Florida
  - The Emory Clinic at Chantilly, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - St. Luke's Cystic Fibrosis Center of Idaho, Boise, Idaho
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - Maine Medical Partners, Portland, Maine
  - Massachusetts General Hospital Cystic Fibrosis Center Clinical Research Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - Harper University Hospital, Detroit, Michigan
  - Spectrum Health Medical Group Adult Cystic Fibrosis Care Center, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Childrens Hospital University of Missouri Health Sciences Center, Columbia, Missouri
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital - St. Louis University, St Louis, Missouri
  - Washington University School of Medicine / St. Louis Children's Hospital, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock, Manchester, New Hampshire
  - Morristown Medical Center, Morristown, New Jersey
  - Albany Medical College, Pulmonary and Critical Care Medicine, Albany, New York
  - CF Therapeutics Development Center of Western New York, Buffalo, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Atrium Health Levine Children's Hospital, Charlotte, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Toledo Children's Hospital/Pediatric Pulmonary & Cystic Fibrosis Center, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Santiago Reyes, M.D., Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Prisma Health Richland Campus, Columbia, South Carolina
  - Sanford Children's Speciality Clinic, Sioux Falls, South Dakota
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nephrology Clinical Trials Center, Nashville, Tennessee
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Health Care System, Fort Worth, Texas
  - Texas Children's Hospital - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Vermont Lung Center, Colchester, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Providence Pediatric Pulmonary & Cystic Fibrosis Clinic, Spokane, Washington
  - West Virginia University, Morgantown, West Virginia
  - University Hospital and UW Health Clinics, Madison, Wisconsin
- Australia (9):
  - Royal Prince Alfred Hospital, Camperdown
  - The Prince Charles Hospital, Chermside
  - Alfred Hospital, Melbourne
  - Institute for Respiratory Health, Nedlands
  - Telethon Kids Institute, Nedlands
  - The Royal Children's Hospital, Parkville
  - Mater Adult Hospital, South Brisbane
  - Queensland Children's Hospital, South Brisbane
  - Westmead Hospital, Westmead
- Austria (4):
  - University of Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Uniklinikum Salzburg - Universitätsklinik für Pneumologie/Lungenheilkunde, Salzburg
  - Medizinische Universität Wien, Vienna
- Belgium (5):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - Universitair Ziekenhuis Brussel - Campus Jette, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- Canada (8):
  - University of Calgary Medical Clinic of the Foothills Medical Centre, Calgary
  - Stollery Children's Hospital, Edmonton
  - St. Joseph's Health Care London, London
  - Centre Hospitalier de l'Universite de Montreal (CHUM) Hotel-Dieu, Montreal
  - McGill University Health Centre, Glen Site, Montreal Children's Hospital, Montreal
  - Institut Universitaire de Cardiologie et Pneumologie de Quebec - Universite Laval, Québec
  - British Columbia Children's Hospital, Vancouver
  - St. Paul's Hospital, Vancouver
- Czechia (2):
  - Klinika Detskych Infekcnich Nemoci, Brno
  - Fakultni nemocnice v Motole, Prague
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Juliane Marie Center, Rigshospitalet, Copenhagen
- France (14):
  - Groupe Hospitaler Pellegrin, CHU De Bordeaux, Bordeaux
  - CHU Lyon - Hopital Femme Mere-Enfant, Bron
  - Centre Hospitalier Intercommunal Creteil, Créteil
  - Institut Cœur Poumon, CHU de Lille, Lille
  - Hopital Arnaud de Villeneuve, Montpellier
  - Centre Hospitalier Universitaire (CHU) de Nice - Hopital Pasteur, Nice
  - Hopital Cochin, Paris
  - Hopital Robert Debre, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre de Perharidy, Roscoff
  - CHU de Rouen - Hopital Charles Nicolle, Rouen
  - Hôpital de Hautepierre, AX5, Strasbourg
  - Hopital Foch (Suresnes), Hopital Foch, Adultes, Suresnes
  - Hopital Bretonneau, Tours
- Germany (14):
  - Charite Paediatric Pulmonology Department, Berlin
  - Friedrich-Alexander University of Erlangen-Nuremberg, University Children's Hospital, Erlangen
  - Kinderklinik III, Abt. fur Pneumologie, Essen
  - Ruhrlandklinik Westdeutsches Lungenzentrum am Klinikum Essen, Essen
  - Johann Wolfgang Goethe University, Frankfurt
  - Justus-Liebig-Universität Gießen Zentrum für Kinderheilkunde und Jugendmedizin, Giessen
  - Hannover Medical School, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Mukoviszidose-Zentrum am Universitätsklinikum Jena, Klinik für Kinder- und Jugendmedizin, Jena
  - Johannes Gutenberg-Universitaet, Mainz
  - Pneumologisches Studienzentrum Muenchen-West, München
  - Klinikum Westbrandenburg (CF), Potsdam
  - Universitätsklinikum Ulm, Klinik für Kinder- und Jugendmedizin (CF), Ulm
  - Universitätsklinikum Würzburg, Würzburg
- Greece (2):
  - General Hospital of Thessaloniki "Papanikolaou", Thessaloniki
  - General Hospital of Thessaloniki 'Hippokratio', 3rd Pediatrics Department of Aristotle University of Thessaloniki, Thessaloniki
- Hungary (2):
  - National Koranyi Institute for TBC and Pulmonology, Budapest
  - Pulmonology Institute Torokbalint, Törökbálint
- Ireland (5):
  - Cork University Hospital, Cork
  - Children's Health Ireland at Crumlin, Dublin
  - Children's Health Ireland at Temple Street, Dublin
  - St. Vincent's University Hospital, Dublin
  - University Hospital Limerick (Pediatrics), Limerick
- Israel (3):
  - Hadassah Medical Organization, Jerusalem
  - Schneider Children's Medical Center of Israel, Petach Tikvah
  - Sheba Medical Center - The Edmond and Lili Safra Children's Hospital, Tel Litwinsky
- Italy (8):
  - Azienda Ospedaliero Universitaria Ospedale Riuniti, Ancona
  - Azienda Ospedaliero Universitaria Ospedale Pediatrico Meyer, Florence
  - IRCCS Istituto Giannina Gaslini-Ospedale Pediatrico, Genova
  - Fondazione IRCCS Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Malattie Apparato Respiratorio 2 - Centro Fibrosi Cistica, Orbassano
  - Centro Regionale Fibrosi Cistica, A.O. Ospedale San Carlo, Potenza
  - Azienda Ospedaliera di Verona - Ospedale Civile Maggiore, Verona
- Netherlands (5):
  - Academisch Medisch Centrum (Academic Medical Centre), Amsterdam
  - UMC St. Radboud, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis van den Haag, The Hague
  - University Medical Center, Utrecht, Department of Pulmonology and Tuberculosis, Utrecht
- New Zealand (4):
  - Canterbury District Health Board, Christchurch
  - Starship Children's Hospital, Grafton
  - Waikato Hospital, Hamilton
  - Greenlane Clinical Centre, One Tree Hill
- Norway (2):
  - Haukeland Universitetssjukehus (CF), Bergen
  - Oslo University Hospital, Department of Paediatric Medicine, Oslo
- Poland (2):
  - Pediatric Hospital Polanki named of Maciej Płażyński, Gdansk
  - Klinika Mukowiscydozy IMD Oddozial Chorob Pluc Szpzoz IM. Dzieci WarszaWY, Łomianki
- Portugal (3):
  - Hospital de Santa Maria, Lisbon
  - CHP - Hospital de Santo Antonio, Porto
  - Hospital Sao Joao, Porto
- Spain (8):
  - Hospital Saint Joan de Deu, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Corporacio Sanitaria Parc Tauli - Sabadell Hospital Universitari, Sabadell
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Lund University Skanes Universitetssjukhus, Lund
  - Karolinska Universitetssjukhuset, Huddinge, Stockholm
- Kinderspital Zuerich, Zurich, Switzerland
- United Kingdom (17):
  - Birmingham Heartlands Hospital, Birmingham
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol Royal Hospital, Bristol
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Western General Hospital, Edinburgh
  - Royal Devon University Healthcare NHS Foundation Trust, Exeter
  - Clinical Research Facility, Queen Elizabeth University Hospital, Glasgow
  - Leeds General Infirmary, Leeds
  - St. James University Hospital, Leeds
  - Liverpool Heart and Chest Hospital, Liverpool
  - King's College Hospital, London
  - Royal Brompton Hospital, London
  - St. Bartholomew's Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Wythenshawe Hospital, Manchester
  - Clinical Research Facility, Newcastle upon Tyne
  - All Wales Adult Cystic Fibrosis Centre, University Hospital Llandough, Penarth
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing